CLINICAL TRIAL: NCT06229327
Title: The Effect of Therapeutic Play on Anxiety and Fear Levels Before Indwelling Catheter Intervention in Children Aged 6-12 Years Followed up in Hematology Oncology Service: a Randomized Controlled Trial
Brief Title: Effects of Therapeutic Play on Anxiety and Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Gülzade Uysal, Associate professor, Okan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0000-0002-4213-175X
Record Dates: First submitted 2023-10-21; First posted 2024-01-29 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEDİATRİC (Experimental): Children in the intervention group were played a therapeutic game explaining the procedure before indwelling catheter intervention. Children in the control group did not undergo any intervention other than the hospital's normal procedure before indwelling catheter intervention.
  Interventions: Behavioral: THERAPEUTICGAMES

INTERVENTIONS:
Behavioral: THERAPEUTICGAMES — THERAPEUTICGAMES

SUMMARY:
This study was carried out as a randomized controlled experimental study in order to evaluate the effect of therapeutic game use on anxiety and fear levels before indwelling catheter intervention in children aged 6-12 years followed in the hematology oncology service. A simple randomization method was used to assign children to groups. Ethics committee and institutional permission was obtained for the research. Research data were obtained from a total of 80 children, 40 interventions and 40 controls, hospitalized in Istanbul Medical Faculty Pediatric Hematology Service between October 2022 and August 2023.

Data; It was evaluated with the information form, child follow-up form, Child Anxiety Scale- State (ÇAS-D) and Child Fear Scale (CCS). For those assigned to the intervention group among the mother and child who signed the informed consent form; Before the indwelling catheter intervention, the children were shown the procedure on the amigrumi knitted baby developed by the researcher, the catheter application area was explained through the cardiovascular image and the catheter to be inserted was shown as an example. For those assigned to the control group; No intervention was applied other than the hospital's normal procedure. Data were evaluated using the SPPS 26 (IBM Corp. IBM 1989, 2019. SPSS Statistics for Windows, Version 26.0. Armonk, NY: IBM Corp.) package program. It was determined that the MCQ and ÇAS-D scores of the children in the intervention group were significantly lower than those in the control group (p˂0.01). It was determined that the mean CTA and respiratory rate of the children in the intervention group just before and 2 hours after the application were lower than the control group (p<0.001).

According to the results of the research, it was determined that the therapeutic game applied before indwelling catheter intervention in children between the ages of 6-12 was effective in reducing children's anxiety and fear.

DETAILED DESCRIPTION:
According to the results of the research, it was determined that the therapeutic game applied before indwelling catheter intervention in children between the ages of 6-12 was effective in reducing children's anxiety and fear.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 6-12 Being diagnosed with cancer Receiving chemotherapy treatment It will be the first time that a permanent catheter will be inserted.

Exclusion Criteria:

* Being in the terminal period Hearing and/or visual impairment Having another health problem or condition that will prevent communication (Turkish inability to speak…etc)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
children's anxiety scores | 30 minutes
  Child Anxiety Scale-Conditioning (min:0-maks:10)
children's fear scores | 30 minutes
  Child Fear Scale (min:0-maks:4)

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Demirer, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Athanassiadou E, Tsiantis J, Christogiorgos S, Kolaitis G. An evaluation of the effectiveness of psychological preparation of children for minor surgery by puppet play and brief mother counseling. Psychother Psychosom. 2009;78(1):62-3. doi: 10.1159/000172623. Epub 2008 Nov 18. No abstract available. PMID 19018160
- [Result] Baranowski T, Blumberg F, Buday R, DeSmet A, Fiellin LE, Green CS, Kato PM, Lu AS, Maloney AE, Mellecker R, Morrill BA, Peng W, Shegog R, Simons M, Staiano AE, Thompson D, Young K. Games for Health for Children-Current Status and Needed Research. Games Health J. 2016 Feb;5(1):1-12. doi: 10.1089/g4h.2015.0026. Epub 2015 Aug 11. PMID 26262772
- [Result] Barton A, Ventura R, Vavrik B. Peripheral intravenous cannulation: protecting patients and nurses. Br J Nurs. 2017 Apr 27;26(8):S28-S33. doi: 10.12968/bjon.2017.26.8.S28. PMID 28453316
- [Result] Bawaeda O, Wanda D, Aprillia Z. Effectiveness of pop-it therapeutic play on children's anxiety during inhalation therapy in children's wards. Pediatr Med Chir. 2023 Mar 28;45(s1). doi: 10.4081/pmc.2023.315. PMID 36974915